CLINICAL TRIAL: NCT07050745
Title: Accelerating Adoption of Patient-centered Cervical Cancer Screening and Treatment Linkage in Kenya
Acronym: DADA-LINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kenyatta National Hospital (Other Government)
Collaborators: Emory University (Other); University of Washington (Other); National Cancer Institute (NCI) (NIH); Kenya Ministry of Health (Other Government); Queen's University (Other); University of Nairobi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P864/11/2023; U54CA284036 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Cervical Cancer Screening; HPV DNA
Keywords: cervical cancer; screening; m-Health; linkage to treatment; VIA; HPV; HPV self-sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A cluster-randomized hybrid type 2 trial will evaluate cervical cancer screening implementation and effectiveness across 20 facilities in Nairobi, Kenya offering primary healthcare. Clinics randomized to the control arm will continue with usual care practices for cervical cancer screening, triage, and treatment. Intervention facilities will provide DADA LINK (HPV self-sampling, care navigators, and mHealth support for cervical cancer screening and treatment linkage).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DADA-LINK Integrated Care Package: HPV Self-Sampling, Care Navigation, and mHealth support (Experimental): Intervention facilities will receive the DADA-LINK multi-component integrated care package comprised of HPV self-sampling, care navigation, and mHealth support.
  Interventions: Behavioral: DADA LINK
- Routine standard of care for cervical cancer screening, linkage and treatment (No Intervention): Clinics randomized to the control arm will continue with usual care practices for cervical cancer screening, triage, and treatment

INTERVENTIONS:
Behavioral: DADA LINK — Intervention facilities will receive the DADA-LINK intervention, comprised of:
  1. HPV self-sampling: We will provide clinics with HPV self-sampling kits to administer to eligible patients.
  2. Care Navigation: One study-supported non-physician care navigator will be assigned to each clinic to support the clinic staff. These trained individuals will be responsible for managing data collection through the mHealth platform to aid the coordination of services and for motivating the clinic staff to adhere to cervical cancer care guidelines.
  3. mHealth support for cervical cancer screening and treatment linkage: The WEMA application is a low-cost and highly adaptable open-source application designed for cervical cancer data monitoring and evaluation. Relevant patient information and data on uptake of cervical cancer screening and triage/treatment will be entered in the WEMA platform. The platform will additionally be used to send text messages to patients to facilitate clinic attendance.
  Arms: DADA-LINK Integrated Care Package: HPV Self-Sampling, Care Navigation, and mHealth support

SUMMARY:
This study aims to test the use of a multi-component care strategy (DADA LINK) designed to improve cervical cancer screening and linkage to treatment. The duration of the trial is 12 months, with a 6-month follow-up period to evaluate intervention costs and measure maintenance of the care strategies. Study staff at each clinic will abstract data on cervical cancer screening and triage/treatment. Clinics randomized to the intervention arm will have care coordinators who motivate clinic staff to adhere to cervical cancer care guidelines, conduct patient exit surveys to assess intervention fidelity, and support care coordination through use of the mHealth platform (WEMA).

DETAILED DESCRIPTION:
The highest global incidence of cervical cancer is in sub-Saharan Africa, and it is the leading cause of cancer mortality among women in Kenya. Barriers to cervical cancer screening and treatment have been identified at the patient-, provider-, and facility-level, demonstrating the need for a multi-strategy approach to enhance cervical cancer control. In this research study, formative qualitative research and clinic mapping processes were conducted with primary care clinics in Nairobi County to select contextually appropriate strategies targeting the primary barriers to cervical cancer screening and linkage to treatment in Nairobi, Kenya. This study seeks to evaluate the implementation and effectiveness of a care package designed to enhance the early detection and treatment of precancerous cervical lesions among women aged 25-49 years in Kenya.

Trained study staff will abstract patient data from existing clinic records to monitor and assess rates of cervical cancer screening and linkage to treatment.

Study staff at the intervention clinics (i.e., care coordinators) will motivate and support clinic staff to adhere to cervical cancer care guidelines. Care coordinators will use a mHealth platform (i.e., WEMA) tailored for use in primary care clinics in Kenya to track patient exit interview responses regarding uptake of HPV self-sampling kits and to support clinic staff by tracking cervical cancer screening, follow-up, and linkage to treatment, when appropriate. WEMA will serve as an information management system in the intervention clinics, providing a data dashboard to track patient follow-up and enable text communication with patients.

ELIGIBILITY:
Inclusion Criteria:

- Women ages 25-49 years

Exclusion Criteria:

* Pregnant women
* Women ≤6 weeks postpartum
* Women already confirmed to have cervical cancer

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1980 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary implementation outcome: Cervical cancer screening uptake | 1 day (on the day of clinic visit)
  Binary endpoint (Yes/No) based on completion of the HPV self-sampling (return of the self-collected HPV swab) or having conducted VIA
Primary effectiveness outcome: Receipt of triage and/or treatment | within 12 months
  Binary endpoint (Yes/No) based on receipt of triage and/or treatment

SECONDARY OUTCOMES:
Secondary effectiveness outcomes: Form of triage and/or treatment received | within 12 months
  Receipt of:
  a) Triage (any next step not exclusively counseling or receipt of results) (yes/no);
Secondary effectiveness outcomes: Form of triage and/or treatment received | within 12 months
  Description: Receipt of: b) Treatment (must be some sort of therapeutic procedure) (yes/no)
Secondary effectiveness outcomes: Form of triage and/or treatment received | within 12 months
  Description: Receipt of: c) Triage and treatment (any next step not exclusively counseling or receipt of results; must be some sort of triage or therapeutic procedure) (yes/no)
Communication of HPV test result to patients via mHealth messages | Within 10 days of results being made available
  Binary endpoint (Yes/No) based on confirmation of HPV test results being sent to the participant's phone via mhealth application (WEMA).

CONTACTS AND LOCATIONS:
Overall Officials: Rose J Kosgei, MBChB,MMed,MSc,Fell.GynOnc,PhD, Principal Investigator — University of Nairobi; Leslie Johnson, MPH, MLitt, PhD, Principal Investigator — Emory University
Locations (1):
- Kenyatta National Hospital, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: At the end of the project
Access Criteria: All IPD submitted as part of the trial publication will be accessible

REFERENCES:
- See also: The DADA LINK project contributes to the BREAKTHROUGH Center by developing a project platform with multidisciplinary expertise that conducts innovative and impactful implementation research focused on closing gaps in cervical cancer continuum in Kenya — https://tree4health.emory.edu/programs/breakthrough.html